CLINICAL TRIAL: NCT05110651
Title: The Danish Pre-HCQ Dialysis Study: Hydroxychloroquine for Prevention of COVID19 in Dialysis-treated Patients With End-stage Renal Disease - A Multicenter Parallel-group Open Randomized Clinical Trial
Brief Title: The Danish Pre-HCQ COVID Dialysis Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding
Sponsor: Nicholas Carlson (Other)
Responsible Party: Sponsor-Investigator, Nicholas Carlson, MD PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D-Pre-HCQ-D104
Record Dates: First submitted 2020-03-29; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: COVID-19; End Stage Renal Disease
MeSH Terms: conditions — COVID-19; Kidney Failure, Chronic | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Multicenter parallel-group open-label randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Active Comparator): Oral hydroxychloroquine 200mg once daily
  Interventions: Drug: Hydroxychloroquine
- No treatment (No Intervention): No treatment

INTERVENTIONS:
Drug: Hydroxychloroquine — Oral Hydroxychloroquine 200mg once daily Dose tapered if blood-hydroxychloroquine levels > 2000ng/ml
  Other Names: Plaquenil
  Arms: Hydroxychloroquine

SUMMARY:
Hydroxychloroquine has been shown to inhibit replication of SARS-CoV-2 in vitro. The presented multicenter parallel-group open-label randomized clinical trial aims to investigate the efficacy of prophylactic hydroxychloroquine on mitigation of risk of hospitalization due to COVID-19 in patients with end-stage renal disease.

DETAILED DESCRIPTION:
The emergence of a novel betacoronavirus designated severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has led to a global pandemic with profound implications for public health. Despite sweeping containment measures, spread of infection is ongoing, with potential ramifications pertaining to availability of health care resources. Preliminary data from Wuhan, China and Northern Italy indicate particular vulnerability of patients >60 years with pre-existing comorbidity leading to increased risk of hospitalization and death. Currently, no specific treatment has demonstrated efficacy against infection with SARS-CoV-2 in a clinical trial. However, chloroquine has been shown to inhibit both viral entry and replication in infection with SARS-CoV-2 in vitro; albeit the specific mechanisms remain unchartered. Chloroquine is an amine acidotropic form of quinine. Previously a first-choice front-line drug for the treatment and prophylaxis of malaria, chloroquine remains one of the most prescribed drugs worldwide. The possible benefit of prophylactic treatment with hydroxychloroquine for mitigation of risk of manifest SARS-COV-2 remains untested. The on-going pandemic entails particular risk for patients on chronic dialysis; chronic dialysis is both associated with profound comorbidity but also requirement of continued ambulant hospital based treatment leading to increased exposure. Consequently, the potential benefit of preventative measures is greatly increased.

Aims and objectives The main objective of the following multicenter parallel-group open-label randomized clinical trial aims to investigate the possible benefit of initiating prophylactic hydroxychloroquine versus no treatment in patients on chronic dialysis for mitigation of risk related to SARS-CoV-2. The anticipated results will provide evidence as to the appropriateness of initiating prophylactic treatment for prevention of symptomatic SARS-CoV-2 in a vulnerable comorbid population with direct and immediate implications for clinical management and public health care beyond renal failure.

Methods A total of 568 dialysis-treated patients with end-stage renal disease will be recruited from all dialysis centers (including satellites) in the Capital region. Patients will be randomized to either oral hydroxychloroquinesulphate 200mg once daily or no treatment for three months. The study is planned as a multicenter, open-label, parallel-group pragmatic randomized clinical study.

Additionally, 100 participants on chronic in-center hemodialysis treatment will be invited to participate in a sub-study focused on SARS-CoV-2 screening and prevention. Patients will undergo screening based on oro-pharyngeal sampling twice weekly. If ≥ 20% of infected patients are identified prior to development of symptoms, results will be applied to advise early SARS-CoV-2 screening in all chronic in-center hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years on chronic dialysis due to end-stage renal disease.
* Competence to understand the study rationale, including potential risks and benefits associated with treatment, necessary for written informed consent.

Exclusion Criteria:

* Prior verified SARS-CoV-2 infection.
* Hypersensitivity reaction to chloroquine, hydroxychloroquine or 4-aminoquinolines
* Electrocardiogram with QTc (Bazett's formula) > 450 ms in males and 460 ms in females
* Patients reliant on digoxin or amiodarone treatment
* Pre-existing psoriasis
* Any pre-existing maculopathy with vision reduction
* Prior sensorineural hearing loss
* Pre-existing severe liver insufficiency (spontaneous international normalized ratio >1.5 within the last year)
* Pre-existing epileptic disease requiring anti-epileptic medication
* Pregnancy or lactation
* Insurmountable Language Barrier
* Participation in other ongoing intervention trials investigating COVID19-related outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-10 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalization due to SARS-CoV-2 infection | 3 months
  Number of patients hospitalized due to COVID-19

SECONDARY OUTCOMES:
SARS-CoV-2 infection | 3 months
  Number of patients with verified SARS-CoV-2 infection
SARS-CoV-2 viral load | 3 months
  SARS-CoV-2 viral count as defined by real-time RNA polymerase chain reaction
All-cause mortality | 3 months
  Number of deaths within the study period
Requirement of mechanical ventilation | 3 months
  Number of patients requiring mechanical ventilation due to SARS-CoV-2 infection within the study period
Admission to intensive care | 3 months
  Number of patients admitted to intensive care due to SARS-CoV-2 infection within the study period

OTHER OUTCOMES:
Duration of hospitalization | 3 months
  Duration in days of hospitalization due to SARS-CoV-2 infection
Duration of mechanical ventilation | 3 months
  Duration in day of mechanical ventilation due to SARS-CoV-2 infection
Duration of admission to intensive care | 3 months
  Duration in days of admission to intensive care due to SARS-CoV-2 infection
Bone marrow suppression | 3 months
  Number of patients with leucopeni < 3000/μL within the study period
Hepatic dysfunction | 3 months
  Number of patients with hepatic dysfunction as defined by an alanine transaminaease > 250U/I within the study period
Cardiac injury | 3 months
  Number of patients with evidence of cardiac injury (creatinine kinase-myocardial band > 5μg/L) within the study period
Sudden cardiac death | 3 months
  Number of patients with sudden cardiac death within the study period
QTc prolongation | 3 months
  Number of patients with QTc prolongation (Bazett's formula; >> 450 ms in males and 460 ms in females)
Positiv SARS-CoV-2 antibody | 3 months
  Number of patients with positive SARS-CoV-2 antibody at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Carlson, MD PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (3):
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - North Zealand Hospital, Hillerød

IPD SHARING:
Plan to Share IPD: Yes
Aggregated de-identified individual participant data for primary and secondary outcomes measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Aggregated data will be available within 12 months of study completion
Access Criteria: All data access requests via email. Requestors will be required to sign a Data Access Agreement